CLINICAL TRIAL: NCT02391779
Title: Flaxseed Lignan Enriched Complex for Blood Pressure Reduction in Elderly Participants With High Normal Blood Pressure or Stage I Hypertension
Brief Title: Flaxseed Lignan Supplementation in Elderly Participants With Stage I Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Jane Alcorn, PhD, University of Saskatchewan
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: FSL132
Record Dates: First submitted 2015-02-28; First posted 2015-03-18 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Hypertension
Keywords: High normal blood pressure; Stage I
MeSH Terms: conditions — Hypertension | interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- BeneFlax® + walking training (Dash) (Experimental): BeneFlax (0.8 g, twice a day) with exercise training (30-60 minutes walking training, 5 times a week) for 8 weeks; all participants encouraged to follow Dash Eating Plan.
  Interventions: Dietary Supplement: BeneFlax®; Behavioral: Walking training; Behavioral: Dash Eating Plan
- Placebo + walking training (Dash) (Placebo Comparator): Placebo (whey powder isocaloric to BeneFlax) with exercise training (30-60 minutes walking training, 5 times a week) for 8 weeks; all participants encouraged to follow Dash Eating Plan.
  Interventions: Behavioral: Walking training; Dietary Supplement: Placebo (Whey Protein); Behavioral: Dash Eating Plan
- BeneFlax® + flexibility training (Dash) (Experimental): BeneFlax (0.8 g, twice a day) with placebo exercise training (flexibility training, 5 times a week) for 8 weeks; all participants encouraged to follow Dash Eating Plan.
  Interventions: Dietary Supplement: BeneFlax®; Behavioral: Flexibility training; Behavioral: Dash Eating Plan
- Placebo + flexibility training (Dash) (Sham Comparator): Placebo (whey powder isocaloric to BeneFlax) with placebo exercise training (flexibility training, 5 times a week) for 8 weeks; all participants encouraged to follow Dash Eating Plan.
  Interventions: Behavioral: Walking training; Behavioral: Flexibility training; Behavioral: Dash Eating Plan

INTERVENTIONS:
Dietary Supplement: BeneFlax® — Daily ingestion of 600 mg SDG/day in 1.6 g SDG-enhanced flax lignan (BeneFlax®) with walking training or flexibility training
  Other Names: Flaxseed lignan enriched complex
  Arms: BeneFlax® + flexibility training (Dash); BeneFlax® + walking training (Dash)
Behavioral: Walking training — 30-60 minutes walking training, 5 days/week.
  Arms: BeneFlax® + walking training (Dash); Placebo + flexibility training (Dash); Placebo + walking training (Dash)
Behavioral: Flexibility training — 5 days/week; e.g. stretching training at home
  Arms: BeneFlax® + flexibility training (Dash); Placebo + flexibility training (Dash)
Dietary Supplement: Placebo (Whey Protein) — 0.6 g/day (an amount equal in volume to BeneFlax®) with walking training or flexibility training
  Arms: Placebo + walking training (Dash)
Behavioral: Dash Eating Plan — Dietary Approaches to Stop Hypertension (DASH), a balanced eating plan - all participants in all treatment arms will be encouraged to adopt a DASH eating plan.

SUMMARY:
Current recommendations today suggest that use of therapeutic lifestyle changes, such as supplementation with specific dietary components and moderate exercise, are appropriate interventions for individuals with borderline high blood pressure. Dietary intervention with natural products, such as flaxseed, is associated with decreased prevalence of cardiovascular disease (Adolphe 2010). Lignans are the active compounds in flaxseed believed to mediate the cardiovascular health benefits following flaxseed consumption (Peterson 2010). Clinical trials indicate benefit of Flax Lignan Enriched Complex (FLC) (BeneFlax® from Archer Daniels Midland, a natural product derived from flaxseed composed of 34-38% lignan) for reducing blood cholesterol and glucose (Pan 2007; Zhang 2008) and blood pressure (Cornish 2009). Furthermore, a recent study in atherosclerosis patients showed significant clinical benefit of flaxseed meal for reducing blood pressure (Rodriguez-Leyva 2013). As a therapeutic lifestyle change that could prevent a need to introduce drug therapy in elderly patients, the effectiveness of FLC supplementation alone or in combination with moderate exercise merits investigation.

ELIGIBILITY:
Inclusion Criteria:

* High normal blood pressure (130/85 - 139/89) or stage I hypertension (140/90 - 150/90)
* Ability to follow simple instructions

Exclusion Criteria:

* Age below 60 years.
* Individuals living in long term care homes.
* Individuals unable to walk for 30 minutes.
* Unstable diabetes, or diabetics taking insulin (note: eligible diabetic participants will undergo additional testing during the study ).
* Current cancer or diagnosed with cancer in the past 2 years.
* Significant liver or other gastrointestinal disorder including inflammatory bowel disease. (While constipation is the most common gastrointestinal problem in the elderly, it would not be a contraindication)
* Significant kidney disorder.
* Have taken oral antibiotics in the past three months
* Unstable or severe cardiac disease, recent myocardial infarction, or stroke (either in past 6 months or significantly affecting physical mobility).
* Unstable other medical disease including, but not limited to, pulmonary disorder, epilepsy and genitourinary disorder.
* Migraine with aura within the last year (as this is a risk factor for stroke).
* Current diagnosis of a bleeding condition, or at risk of bleeding.
* Significant immune-compromise.
* Current use of hormone replacement therapy (except thyroid).
* Current use of blood pressure medications and/or diuretics
* Current use of flax seed supplement
* Participation in any other clinical trial with an investigational agent within one month prior to randomization.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in 24 h ambulatory systolic blood pressure | Baseline, week 4, and week 8
  Reduction in 24 h ambulatory systolic blood pressure at midpoint (week 4) and end (week 8) of the intervention relative to baseline value is the primary outcome of the intervention.

SECONDARY OUTCOMES:
Change in body weight | Baseline, week 4, and week 8
  Change in body weight at midpoint (week 4) and end (week 8) of the intervention relative to baseline value.
Heart rate | Baseline
Glucometer fasting blood glucose | Baseline
  Diabetes only; Blood glucose monitored to ensure intervention does not result in hypoglycemia.
Change in blood markers of safety and cardiovascular disease risk factors (clinical biochemical panel including fasting glucose, lipids, cholesterol, electrolytes, C-reactive protein) | Baseline, week 4, and week 8
  These parameters will be measured individual but reviewed as a composite to confirm safety and any change in cardiovascular disease risk.
Blood levels of the flax lignan, secoisolariciresinol diglucoside (SDG), and its metabolites | Week 4
Physical activity assessment tool (PASE) | Baseline
Block Food Frequency Questionnaire | Baseline
Change in Body composition by DXA (Dual-energy X-ray absorptiometry) | Baseline, week 4, and week 8
  Change in body composition at midpoint (week 4) and end (week 8) of the intervention relative to baseline value.
Heart Rate | week 4
Heart Rate | Week 8
Change in lying and standing blood pressure | Baseline, week 4, and week 8
  Change in lying and standing blood pressure at midpoint (week 4) and end (week 8) of the intervention relative to baseline value.
Respiratory rate | Baseline
Respiratory rate | Week 4
Respiratory rate | Week 8
Block Food Frequency Questionnaire | Week 8
Blood levels of the flax lignan, secoisolariciresinol diglucoside (SDG), and its metabolites | Week 8
Glucometer fasting blood glucose | Week 4
  Diabetes only; Blood glucose monitored to ensure intervention does not result in hypoglycemia.
Glucometer fasting blood glucose | Week 8
  Diabetes only; Blood glucose monitored to ensure intervention does not result in hypoglycemia.

OTHER OUTCOMES:
Number of participants with adverse events as a safety measurement | Continuously throughout 9 weeks
Number of participants with severe non-compliance with the protocol | Continuously throughout 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jane Alcorn, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- College of Pharmacy, University of Saskatchewan, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Background] Peterson J, Dwyer J, Adlercreutz H, Scalbert A, Jacques P, McCullough ML. Dietary lignans: physiology and potential for cardiovascular disease risk reduction. Nutr Rev. 2010 Oct;68(10):571-603. doi: 10.1111/j.1753-4887.2010.00319.x. PMID 20883417
- [Background] Pan A, Sun J, Chen Y, Ye X, Li H, Yu Z, Wang Y, Gu W, Zhang X, Chen X, Demark-Wahnefried W, Liu Y, Lin X. Effects of a flaxseed-derived lignan supplement in type 2 diabetic patients: a randomized, double-blind, cross-over trial. PLoS One. 2007 Nov 7;2(11):e1148. doi: 10.1371/journal.pone.0001148. PMID 17987126
- [Background] Zhang W, Wang X, Liu Y, Tian H, Flickinger B, Empie MW, Sun SZ. Dietary flaxseed lignan extract lowers plasma cholesterol and glucose concentrations in hypercholesterolaemic subjects. Br J Nutr. 2008 Jun;99(6):1301-9. doi: 10.1017/S0007114507871649. Epub 2007 Dec 6. PMID 18053310
- [Background] Cornish SM, Chilibeck PD, Paus-Jennsen L, Biem HJ, Khozani T, Senanayake V, Vatanparast H, Little JP, Whiting SJ, Pahwa P. A randomized controlled trial of the effects of flaxseed lignan complex on metabolic syndrome composite score and bone mineral in older adults. Appl Physiol Nutr Metab. 2009 Apr;34(2):89-98. doi: 10.1139/H08-142. PMID 19370038
- [Background] Rodriguez-Leyva D, Weighell W, Edel AL, LaVallee R, Dibrov E, Pinneker R, Maddaford TG, Ramjiawan B, Aliani M, Guzman R, Pierce GN. Potent antihypertensive action of dietary flaxseed in hypertensive patients. Hypertension. 2013 Dec;62(6):1081-9. doi: 10.1161/HYPERTENSIONAHA.113.02094. Epub 2013 Oct 14. PMID 24126178
- [Background] Adolphe JL, Whiting SJ, Juurlink BH, Thorpe LU, Alcorn J. Health effects with consumption of the flax lignan secoisolariciresinol diglucoside. Br J Nutr. 2010 Apr;103(7):929-38. doi: 10.1017/S0007114509992753. Epub 2009 Dec 15. PMID 20003621